CLINICAL TRIAL: NCT02594124
Title: An Open-Label Extension Study for Patients With Spinal Muscular Atrophy Who Previously Participated in Investigational Studies of ISIS 396443
Brief Title: A Study for Participants With Spinal Muscular Atrophy (SMA) Who Previously Participated in Nusinersen (ISIS 396443) Investigational Studies
Acronym: SHINE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ISIS 396443-CS11; 2015-001870-16 (EudraCT Number)
Expanded Access: NCT02865109 (No longer available)
Record Dates: First submitted 2015-10-30; First posted 2015-11-02 (Estimated); Results first posted 2024-10-22 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-09

CONDITIONS: Spinal Muscular Atrophy
Keywords: SMA; SMN; SMNRx; ISIS-SMNRx; ISIS 396443; SHINE; IONIS-SMNRx; IONIS-SMN Rx; Spinraza; nusinersen
MeSH Terms: conditions — Muscular Atrophy, Spinal | interventions — nusinersen

STUDY DESIGN:
Masking Description: During the blinded loading period, the following participants will be masked:
  * Key site personnel (Investigator, Study Coordinator, and Outcomes Assessors)
  * Participant
  * The sponsor
  After the loading period has been completed, subsequent doses will be unblinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (5):
- Group 1 (Experimental): Participants transitioned from ISIS 396443-CS3B (NCT02193074)
  Interventions: Drug: nusinersen
- Group 2 (Experimental): Participants transitioned from ISIS 396443-CS4 (NCT02292537)
  Interventions: Drug: nusinersen
- Group 3 (Experimental): Participants transitioned from ISIS 396443-CS12 (NCT02052791)
  Interventions: Drug: nusinersen
- Group 4 (Experimental): Participants transitioned from ISIS 396443-CS3A (NCT01839656)
  Interventions: Drug: nusinersen
- Group 5 (Experimental): Participants transitioned from 232SM202 (NCT02462759)
  Interventions: Drug: nusinersen

INTERVENTIONS:
Drug: nusinersen — Administered by intrathecal (IT) injection
  Other Names: ISIS 396443; Spinraza; BIIB058; IONIS SMN Rx; ISIS SMNRx

SUMMARY:
The primary objective is to evaluate long-term safety and tolerability of nusinersen (ISIS 396443) administered by intrathecal (IT) injection to participants with Spinal Muscular Atrophy (SMA) who previously participated in investigational studies of nusinersen. The secondary objective is to examine the long-term efficacy of nusinersen administered by IT injection to participants with SMA who previously participated in investigational studies of nusinersen.

DETAILED DESCRIPTION:
This study was initiated and the protocol was registered by Ionis Pharmaceuticals, Inc.

In August 2016, Biogen assumed responsibility for this study.

ELIGIBILITY:
Key Inclusion Criteria:

* Signed informed consent of parent or guardian and signed informed assent of participant, if indicated per participant's age and institutional guidelines.
* Completion of the index study in accordance with the study protocol or as a result of Sponsor decision (e.g., early termination of the index study) within the preceding 16 weeks

Key Exclusion Criteria:

* Have any condition or worsening condition which in the opinion of the Investigator would make the participant unsuitable for enrollment, or could interfere with the participant participating in or completing the study
* Clinically significant abnormalities in hematology or clinical chemistry parameters or electrocardiogram (ECG), as assessed by the Site Investigator, at the Screening visit that would render the participant unsuitable for participation in the study
* Participant's parent or legal guardian is not willing or able to meet standard of care guidelines (including vaccinations and respiratory syncytial virus prophylaxis if available), nor provide nutritional and respiratory support throughout the study
* Treatment with another investigational agent, biological agent, or device within one month of Screening, or 5 half-lives of study agent, whichever is longer

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 292 (Actual)
Dates: Start 2015-11-04 (Actual); Primary Completion 2023-08-21 (Actual); Study Completion 2023-08-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (47):
- United States (18):
  - David Geffen School of Medicine at UCLA, Los Angeles, California
  - Stanford University School of Medicine, Palo Alto, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Nemours Children's Clinic, Orlando, Florida
  - Ann & Robert H. Lurie Children's Hospital of Chicago, New York, Illinois
  - The Johns Hopkins Hospital, Baltimore, Maryland
  - Boston Children's Hospital, Boston, Massachusetts
  - Gillette Children's Specialty Healthcare, Saint Paul, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Columbia University Medical Center, New York, New York
  - Duke University School of Medicine, Durham, North Carolina
  - Duke University School of Medicine, Miyagi, North Carolina
  - Oregon Health Sciences University, Durham, Oregon
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Medical Center, Dallas, Texas
  - University of Utah, Obu, Aichi, Utah
  - Seattle Children's Hospital, Seattle, Washington
- Australia (2):
  - Sydney Children's Hospital Clinical Research Centre, Sydney, New South Wales
  - Royal Children's Hospital, Parkville, Victoria
- Universitair Kinderziekenhuis Koningin Fabiola, Brussels, Belgium
- Canada (3):
  - BC Children's Hospital / UBC, Vancouver, British Columbia
  - Children's Health Research Institute, Brussel, Ontario
  - McGill University Health Centre, Montreal, Quebec
- Armand Trousseau Hospital, I-Motion, Paris, Paris 9, France
- Germany (3):
  - LMU-Campus Innenstadt, Munich, Bavaria
  - Universitatsklinikum Essen, Essen
  - Universitaetsklinikum Freiburg, Freiburg im Breisgau
- The University of Hong Kong, Hong Kong, Hong Kong SAR, Hong Kong
- Italy (3):
  - Pediatric Neurology Unit, Catholic University, Essen
  - Istituto Giannina Gaslini, Centro Traslazionale di Miologia, Genova
  - Department of Neuroscience, Università di Messina, AOU Polic, Messina
- Japan (6):
  - Aichi Children's Health and Medical Center, Ōbu, Aichi-ken
  - Hyogo College of Medicine, Nishinomiya, Hyōgo
  - Tokyo Women's Medical University, Shinjuku-ku, Tokyo
  - Kumamoto University Hospital, Kumamoto
  - Miyagi Prefectural Children Hospital, Miyagi
  - University of Miyazaki Hospital, Miyazaki
- Seoul National University Hospital, Seoul, Korea, South Korea
- Spain (3):
  - Hospital Sant Joan de Deu, Barcelona
  - Hospital Universitario Vall de Hebron, Hebron
  - Hospital Universitario La Paz, Madrid
- The Queen Silvia Children's Hospital, Gothenburg, Sweden
- Turkey (Türkiye) (2):
  - Uníversity of Hacettepe, Ankara
  - Marmara University Pendik Training and Research Hospital, Istanbul
- United Kingdom (2):
  - MRC Centre for Neuromuscular Diseases at Newcastle, Newcastle, Northumberland
  - UCL Institute of Child Health, London

REFERENCES:
- See also: Cure SMA — http://www.curesma.org
- See also: Muscular Dystrophy Association — http://mda.org/disease/spinal-muscular-atrophy
- See also: National Organization for Rare Diseases — https://www.rarediseases.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at the investigative sites in Australia, Belgium, Canada, Germany, Spain, France, United Kingdom, Hong Kong, Italy, Japan, Republic of Korea, Sweden, Turkey, and the United States from 04 November 2015 to 21 August 2023.
Pre-assignment Details: A total of 292 participants with infantile and later onset spinal muscular atrophy (SMA) who previously participated in ISIS 396443-CS3B[NCT02193074], ISIS 396443-CS4[NCT02292537], ISIS 396443-CS3A[NCT01839656], ISIS 396443-CS12[NCT02052791] and 232SM202[NCT02462759] were enrolled and treated in this study.
Groups:
- Infantile SMA Onset CS3A: Participants who received nusinersen in study ISIS 396443-CS3A, in an open-label period, received maintenance doses of nusinersen, intrathecal (IT) injection, on days 1, 120, 240, 360, 480, 600, 720, 840, 960, 1080, 1200, 1320, 1440, 1560, and 1680 in Modified Maintenance Dosing Regimen (MMDR) period of this study.
- Infantile SMA Onset CS3B Previous Control: Participants who received sham procedures in study ISIS 396443-CS3B, in a double-blind period, received 4 loading doses of nusinersen IT injection on Days 1, 15, 29, and 64 followed by maintenance doses of nusinersen IT injection, on days 1, 120, 240, 360, 480, 600, 720, 840, 960, 1080, 1200, 1320, 1440, 1560, and 1680 in MMDR period of this study.
- Infantile SMA Onset CS3B Previous ISIS 396443: Participants who received nusinersen in study ISIS 396443-CS3B, in the double-blind period, received 3 sham procedures on Days 1, 15, and 64 and 1 loading dose of nusinersen IT injection on Day 29 followed by maintenance doses of nusinersen IT injection, on days 1, 120, 240, 360, 480, 600, 720, 840, 960, 1080, 1200, 1320, 1440, 1560, and 1680 in MMDR period of this study.
- Infantile SMA Onset 232SM202; Later SMA Onset 232SM202: Participants who received nusinersen in study 232SM202 (i.e., Part 2) in an open-label period, received maintenance doses of nusinersen IT injection, on days 1, 120, 240, 360, 480, 600, 720, 840, 960, 1080, 1200, 1320, 1440, 1560, and 1680 in MMDR period of this study.
- Later SMA Onset CS12 Type 2; Later SMA Onset CS12 Type 3: Participants who received nusinersen in study ISIS 396443-CS12 in an open-label period, received maintenance doses of nusinersen IT injection, on days 1, 120, 240, 360, 480, 600, 720, 840, 960, 1080, 1200, 1320, 1440, 1560, and 1680 in MMDR period of this study.
- Later SMA Onset CS4 Previous Control: Participants who received sham procedures in the study ISIS 396443-CS4 in a double-blind period received 3 loading doses of nusinersen administered by IT injection on Days 1, 29, and 85 followed by maintenance doses of nusinersen IT injection, on days 1, 120, 240, 360, 480, 600, 720, 840, 960, 1080, 1200, 1320, 1440, 1560, and 1680 in MMDR period of this study.
- Later SMA Onset CS4 Previous ISIS 396443: Participants who received nusinersen in the study ISIS 396443-CS4 in a double-blind period received 2 loading doses of nusinersen administered by IT injection on Days 1 and 85 and 1 sham procedure on Day 29 followed by maintenance doses of nusinersen IT injection, on days 1, 120, 240, 360, 480, 600, 720, 840, 960, 1080, 1200, 1320, 1440, 1560, and 1680 in MMDR period of this study.
Period: Overall Study
Arm/Group | Infantile SMA Onset CS3A | Infantile SMA Onset CS3B Previous Control | Infantile SMA Onset CS3B Previous ISIS 396443 | Infantile SMA Onset 232SM202 | Later SMA Onset CS12 Type 2 | Later SMA Onset CS12 Type 3 | Later SMA Onset CS4 Previous Control | Later SMA Onset CS4 Previous ISIS 396443 | Later SMA Onset 232SM202
Started | 13 | 24 | 65 | 12 | 20 | 25 | 42 | 83 | 8
Completed | 10 | 10 | 42 | 7 | 12 | 20 | 19 | 44 | 5
Not Completed | 3 | 14 | 23 | 5 | 8 | 5 | 23 | 39 | 3
Not completed — Adverse Event | 0 | 5 | 8 | 1 | 0 | 0 | 2 | 2 | 0
Not completed — Withdrawal by Subject | 2 | 3 | 5 | 1 | 8 | 4 | 13 | 19 | 0
Not completed — Physician Decision | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Commercial drug | 0 | 1 | 6 | 3 | 0 | 0 | 7 | 11 | 2
Not completed — Reason Not Specified | 1 | 3 | 4 | 0 | 0 | 1 | 1 | 6 | 1

BASELINE CHARACTERISTICS:
Population: The safety analysis set included all participants who were enrolled and received at least 1 dose of nusinersen or underwent sham procedure during CS11.
Groups:
- Infantile SMA Onset CS3A: Participants who received nusinersen in study ISIS 396443-CS3A, in an open-label period, received maintenance doses of nusinersen, IT injection, on days 1, 120, 240, 360, 480, 600, 720, 840, 960, 1080, 1200, 1320, 1440, 1560, and 1680 in MMDR period of this study.
- Total: Total of all reporting groups
Arm/Group | Infantile SMA Onset CS3A | Infantile SMA Onset CS3B Previous Control | Infantile SMA Onset CS3B Previous ISIS 396443 | Infantile SMA Onset 232SM202 | Later SMA Onset CS12 Type 2 | Later SMA Onset CS12 Type 3 | Later SMA Onset CS4 Previous Control | Later SMA Onset CS4 Previous ISIS 396443 | Later SMA Onset 232SM202 | Total
Number analyzed (Participants) | 13 | 24 | 65 | 12 | 20 | 25 | 42 | 83 | 8 | 292
Age, Customized [Count of Participants; unit: Participants]
  Infants and toddlers (28 days-23 months) | 0 | 24 | 65 | 0 | 0 | 0 | 0 | 0 | 0 | 89
  Children (2-11 years) | 13 | 0 | 0 | 12 | 19 | 10 | 42 | 83 | 8 | 187
  Adolescents (12-17 years) | 0 | 0 | 0 | 0 | 0 | 12 | 0 | 0 | 0 | 12
  Adults (18-64 years) | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 0 | 0 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 15 | 36 | 6 | 8 | 15 | 21 | 46 | 3 | 156
  Male | 7 | 9 | 29 | 6 | 12 | 10 | 21 | 37 | 5 | 136
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 3 | 10 | 2 | 2 | 6 | 0 | 4 | 1 | 29
  Not Hispanic or Latino | 12 | 18 | 47 | 7 | 18 | 19 | 37 | 69 | 5 | 232
  Unknown or Not Reported | 0 | 3 | 8 | 3 | 0 | 0 | 5 | 10 | 2 | 31
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 2
  Asian | 1 | 1 | 2 | 4 | 1 | 1 | 7 | 16 | 0 | 33
  Black or African American | 0 | 0 | 3 | 0 | 0 | 1 | 1 | 1 | 0 | 6
  White | 10 | 18 | 47 | 5 | 18 | 23 | 26 | 53 | 4 | 204
  Multiple | 1 | 2 | 1 | 0 | 1 | 0 | 3 | 3 | 0 | 11
  Other | 1 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 1 | 5
  Not reported | 0 | 3 | 8 | 3 | 0 | 0 | 5 | 10 | 2 | 31

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: AE:unfavorable and unintended sign, symptom, or disease temporally associated with study/use of an investigational drug, whether or not it's considered related to investigational drug. SAE:AE that in view of either Investigator/Sponsor, meets any of the following criteria: results in death;is life-threatening:i.e.poses risk of death, hospitalization/it's prolongation;results in a persistent or significant incapacity or substantial disruption of normal life functions;results in congenital anomaly or birth defect in offspring;is an important event in the opinion of Investigator/Sponsor. TEAE: if it was present prior to first dose of nusinersen or first sham procedure in index study and subsequently worsened in severity/was not present prior to first dose of nusinersen or first sham procedure in index study but subsequently appeared.
Time Frame: From Day 1 up to the end of the study (up to 2848 days)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Infantile SMA Onset CS3A | Infantile SMA Onset CS3B Previous Control | Infantile SMA Onset CS3B Previous ISIS 396443 | Infantile SMA Onset 232SM202 | Later SMA Onset CS12 Type 2 | Later SMA Onset CS12 Type 3 | Later SMA Onset CS4 Previous Control | Later SMA Onset CS4 Previous ISIS 396443 | Later SMA Onset 232SM202
Number analyzed (Participants) | 13 | 24 | 65 | 12 | 20 | 25 | 42 | 83 | 8
Participants
  AEs | 13 | 24 | 65 | 12 | 20 | 25 | 42 | 80 | 8
  SAEs | 11 | 23 | 59 | 9 | 12 | 6 | 26 | 47 | 5

2. Primary Outcome: Number of Participants With Vital Sign Abnormalities Reported as AEs
Description: The vital sign assessments included blood pressure, temperature, pulse rate, and respiratory rate. Participants with abnormalities in these assessments recorded as AEs were reported.
Time Frame: From Day 1 up to the end of the study (up to 2848 days)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Infantile SMA Onset CS3A | Infantile SMA Onset CS3B Previous Control | Infantile SMA Onset CS3B Previous ISIS 396443 | Infantile SMA Onset 232SM202 | Later SMA Onset CS12 Type 2 | Later SMA Onset CS12 Type 3 | Later SMA Onset CS4 Previous Control | Later SMA Onset CS4 Previous ISIS 396443 | Later SMA Onset 232SM202
Number analyzed (Participants) | 13 | 24 | 65 | 12 | 20 | 25 | 42 | 83 | 8
Participants
  Bradycardia | 1 | 0 | 6 | 1 | 0 | 0 | 1 | 0 | 0
  Tachycardia | 2 | 4 | 5 | 1 | 0 | 0 | 1 | 2 | 0
  Pyrexia | 13 | 15 | 50 | 5 | 10 | 3 | 21 | 39 | 5
  Body Temperature Increased | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0
  Heart Rate Increased | 3 | 2 | 4 | 3 | 0 | 0 | 2 | 0 | 0
  Oxygen Saturation Decreased | 1 | 9 | 20 | 2 | 0 | 1 | 2 | 3 | 0
  Respiratory Rate Increased | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Tachypnoea | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0

3. Primary Outcome: Number of Participants With Weight Abnormalities Reported as AEs
Description: Weight decrease was characterized by a decrease of >=7% from baseline and weight increase was characterized by an increase of >=7% from baseline. Participants with these abnormalities recorded as AEs were reported.
Time Frame: From Day 1 up to the end of the study (up to 2848 days)
Population: The safety analysis set included all participants who were enrolled and received at least 1 dose of nusinersen or underwent sham procedure during CS11. '
Measure: Count of Participants; unit: Participants
Arm/Group | Infantile SMA Onset CS3A | Infantile SMA Onset CS3B Previous Control | Infantile SMA Onset CS3B Previous ISIS 396443 | Infantile SMA Onset 232SM202 | Later SMA Onset CS12 Type 2 | Later SMA Onset CS12 Type 3 | Later SMA Onset CS4 Previous Control | Later SMA Onset CS4 Previous ISIS 396443 | Later SMA Onset 232SM202
Number analyzed (Participants) | 13 | 24 | 65 | 12 | 20 | 25 | 42 | 83 | 8
Participants
  Weight Decreased | 0 | 0 | 3 | 1 | 0 | 1 | 1 | 3 | 0
  Weight Increased | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 0 | 0

4. Primary Outcome: Number of Participants With Neurological Abnormalities Reported as AEs
Description: Participants with abnormalities in neurological examinations recorded as AEs were reported.
Time Frame: From Day 1 up to the end of the study (up to 2848 days)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Infantile SMA Onset CS3A | Infantile SMA Onset CS3B Previous Control | Infantile SMA Onset CS3B Previous ISIS 396443 | Infantile SMA Onset 232SM202 | Later SMA Onset CS12 Type 2 | Later SMA Onset CS12 Type 3 | Later SMA Onset CS4 Previous Control | Later SMA Onset CS4 Previous ISIS 396443 | Later SMA Onset 232SM202
Number analyzed (Participants) | 13 | 24 | 65 | 12 | 20 | 25 | 42 | 83 | 8
Participants
  Areflexia | 2 | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 0
  Hyporeflexia | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Nystagmus | 0 | 0 | 4 | 1 | 0 | 0 | 0 | 0 | 0
  Motor Dysfunction | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Muscle Contractions Involuntary | 0 | 0 | 0 | 1 | 2 | 1 | 1 | 4 | 0
  Myoclonus | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Paraesthesia | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1
  Tremor | 1 | 0 | 1 | 0 | 1 | 1 | 1 | 3 | 0

5. Primary Outcome: Number of Participants With Laboratory Abnormalities Reported as AEs
Description: Laboratory investigations included hematology, coagulation, serum chemistry and urinalysis parameters. Participants with abnormalities in these laboratory investigations recorded as AEs were reported.
Time Frame: From Day 1 up to the end of the study (up to 2848 days)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Infantile SMA Onset CS3A | Infantile SMA Onset CS3B Previous Control | Infantile SMA Onset CS3B Previous ISIS 396443 | Infantile SMA Onset 232SM202 | Later SMA Onset CS12 Type 2 | Later SMA Onset CS12 Type 3 | Later SMA Onset CS4 Previous Control | Later SMA Onset CS4 Previous ISIS 396443 | Later SMA Onset 232SM202
Number analyzed (Participants) | 13 | 24 | 65 | 12 | 20 | 25 | 42 | 83 | 8
Participants
  Anaemia | 1 | 0 | 6 | 1 | 2 | 0 | 1 | 1 | 1
  Leukocytosis | 1 | 0 | 3 | 0 | 0 | 0 | 1 | 2 | 0
  Leukopenia | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Lymphopenia | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Neutropenia | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
  Neutrophilia | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 2 | 0
  Pancytopenia | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Thrombocytopenia | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
  Thrombocytosis | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Hypertransaminasaemia | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
  Pyuria | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Urinary Tract Infection | 3 | 3 | 11 | 1 | 2 | 1 | 4 | 7 | 1
  Alanine Aminotransferase Increased | 0 | 1 | 3 | 0 | 0 | 0 | 0 | 1 | 0
  Aspartate Aminotransferase Increased | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0
  Blood Albumin Decreased | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Blood Bicarbonate Decreased | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
  Blood Calcium Decreased | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Blood Osmolarity Increased | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Blood Potassium Abnormal | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Blood Potassium Decreased | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Blood Potassium Increased | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Crystal Urine Present | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 6 | 0
  Full Blood Count Decreased | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Full Blood Count Increased | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Gamma-Glutamyltransferase Increased | 0 | 2 | 3 | 0 | 0 | 0 | 0 | 0 | 0
  Haemoglobin Decreased | 0 | 1 | 2 | 1 | 0 | 0 | 0 | 0 | 0
  Hepatic Enzyme Increased | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0
  Liver Function Test Increased | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Mean Platelet Volume Decreased | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Neutrophil Count Decreased | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Neutrophil Count Increased | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Platelet Count Decreased | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
  Platelet Count Increased | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Protein Urine Present | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 3 | 0
  Red Blood Cell Count Increased | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Transaminases Increased | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Urine Ketone Body Present | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  White Blood Cell Count Increased | 0 | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 0
  White Blood Cells Urine | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  White Blood Cells Urine Positive | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
  Hypercalcaemia | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Hyperglycaemia | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
  Hypernatraemia | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 1 | 0
  Hypoalbuminaemia | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Hypocalcaemia | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Hypochloraemia | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
  Hypoglycaemia | 2 | 0 | 5 | 0 | 0 | 0 | 1 | 2 | 0
  Hypokalaemia | 1 | 3 | 10 | 0 | 0 | 0 | 1 | 2 | 0
  Hyponatraemia | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 1 | 0
  Electrolyte Imbalance | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0
  Bilirubinuria | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Haematuria | 1 | 1 | 0 | 0 | 0 | 1 | 1 | 2 | 0
  Ketonuria | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Leukocyturia | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0
  Proteinuria | 0 | 1 | 7 | 1 | 0 | 2 | 2 | 8 | 0
  Bandaemia | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0

6. Primary Outcome: Number of Participants With Coagulation Parameters Reported as AEs
Description: Coagulation parameters included activated partial thromboplastin time (aPTT) and international normalized ratio (INR). Participants with abnormalities in these coagulation parameters recorded as AEs were reported.
Time Frame: From Day 1 up to the end of the study (up to 2848 days)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Groups:
- Later SMA Onset 232SM202: Participants entering the study after receiving nusinersen during the open-label phase of Study 232SM202 (i.e., Part 2) received maintenance doses of nusinersen approximately every 4 months according to the MMDR dosing schedule.
Arm/Group | Infantile SMA Onset CS3A | Infantile SMA Onset CS3B Previous Control | Infantile SMA Onset CS3B Previous ISIS 396443 | Infantile SMA Onset 232SM202 | Later SMA Onset CS12 Type 2 | Later SMA Onset CS12 Type 3 | Later SMA Onset CS4 Previous Control | Later SMA Onset CS4 Previous ISIS 396443 | Later SMA Onset 232SM202
Number analyzed (Participants) | 13 | 24 | 65 | 12 | 20 | 25 | 42 | 83 | 8
Participants
  Activated Partial Thromboplastin Time Prolonged | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0
  International Normalised Ratio Abnormal | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  International Normalised Ratio Decreased | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Coagulopathy | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0

7. Primary Outcome: Number of Participants With Clinically Significant Shifts in12 Lead Electrocardiogram (ECG) Results
Description: Clinical significance of abnormalities in 12 lead ECG was determined based on the investigator's discretion.
Time Frame: From Day 1 up to the end of the study (up to 2848 days)
Population: The safety analysis set included all participants who were enrolled and received at least 1 dose of nusinersen or underwent sham procedure during CS11. 'Number analyzed' signifies number of participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Infantile SMA Onset CS3A | Infantile SMA Onset CS3B Previous Control | Infantile SMA Onset CS3B Previous ISIS 396443 | Infantile SMA Onset 232SM202 | Later SMA Onset CS12 Type 2 | Later SMA Onset CS12 Type 3 | Later SMA Onset CS4 Previous Control | Later SMA Onset CS4 Previous ISIS 396443 | Later SMA Onset 232SM202
Number analyzed (Participants) | 13 | 24 | 65 | 12 | 20 | 25 | 42 | 83 | 8
Participants | 2 | 1 | 6 | 1 | 0 | 0 | 1 | 1 | 0

8. Primary Outcome: Number of Participants Taking Any Concomitant Medication
Description: A concomitant therapy is any non-protocol-specified drug or substance (including over-the-counter medications, herbal medications, and vitamin supplements) administered between the beginning of screening and the last telephone contact or study visit.
Time Frame: From Day 1 up to the end of the study (up to 2848 days)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Infantile SMA Onset CS3A | Infantile SMA Onset CS3B Previous Control | Infantile SMA Onset CS3B Previous ISIS 396443 | Infantile SMA Onset 232SM202 | Later SMA Onset CS12 Type 2 | Later SMA Onset CS12 Type 3 | Later SMA Onset CS4 Previous Control | Later SMA Onset CS4 Previous ISIS 396443 | Later SMA Onset 232SM202
Number analyzed (Participants) | 13 | 24 | 65 | 12 | 20 | 25 | 42 | 83 | 8
Participants | 13 | 24 | 65 | 12 | 20 | 25 | 42 | 83 | 8

9. Secondary Outcome: Mean Number of New Motor Milestones Achieved as Assessed by World Health Organization (WHO) Criteria
Description: The WHO motor milestones are a set of six milestones in motor development, all of which would be expected to be attained by 24 months of age in healthy children. The individual milestones are: sitting without support, standing with assistance, hands and knees crawling, walking with assistance, standing alone and walking alone. Mean of number of new milestones achieved was calculated and reported in this outcome measure.
Time Frame: MMDR Period: At Day 1800
Population: The safety analysis set included all participants who were enrolled and received at least 1 dose of nusinersen or underwent sham procedure during CS11. 'Overall number of participants analyzed' signifies number of participants with data available for outcome measure analysis.
Measure: Mean (Standard Deviation); unit: motor milestone
Arm/Group | Infantile SMA Onset CS3A | Infantile SMA Onset CS3B Previous Control | Infantile SMA Onset CS3B Previous ISIS 396443 | Infantile SMA Onset 232SM202 | Later SMA Onset CS12 Type 2 | Later SMA Onset CS12 Type 3 | Later SMA Onset CS4 Previous Control | Later SMA Onset CS4 Previous ISIS 396443 | Later SMA Onset 232SM202
Number analyzed (Participants) | 9 | 10 | 43 | 8 | 12 | 18 | 19 | 45 | 6
motor milestone | 0.4 (0.73) | 0.0 (0.00) | 0.7 (1.15) | 0.0 (0.53) | -0.6 (0.79) | -0.1 (0.73) | -0.1 (0.32) | -0.2 (0.60) | -0.2 (0.75)

10. Secondary Outcome: Percentage of Participants With <2 Years of Age Who Attained Motor Milestones as Assessed by Section 2 of Hammersmith Infant Neurological Examination (HINE)
Description: HINE is evaluated in infants between 2-24 months of age. It's a simple, standardized instrument including 26 items assessing different aspects of neurological examinations, such as cranial nerves, posture, movements, tone, and reflexes. In this study, Module 2 of HINE (HINE-2) was assessed, which evaluates 8 developmental milestones (head control, sitting, voluntary grasp, ability to kick, rolling, crawling, standing, and walking) scored on a 3, 4, or 5-point scale, with 0 indicating inability to perform task and score of 2, 3, or 4 indicating full milestone development. Total score is calculated by summing item scores to give maximum possible score of 26. Higher score indicates good neurological function.
Time Frame: At Day 309
Population: The safety analysis set included all participants who were enrolled and received at least 1 dose of nusinersen or underwent sham procedure during CS11. 'Overall number of participants analyzed' signifies number of participants with data available for outcome measure analysis. Only CS3A and CS3B arm groups were planned to be analyzed for this outcome measure (OM).
Measure: Number; unit: percentage of participants
Arm/Group | Infantile SMA Onset CS3A | Infantile SMA Onset CS3B Previous Control | Infantile SMA Onset CS3B Previous ISIS 396443
Number analyzed (Participants) | 8 | 22 | 62
percentage of participants
  Head Control: Unable to Maintain Head Upright | 13 | 86 | 34
  Head Control: Wobbles | 13 | 9 | 18
  Head Control: All the Time Maintained Upright | 75 | 5 | 48
  Sitting: Cannot Sit | 13 | 100 | 39
  Sits With Support at Hips | 13 | 0 | 19
  Sitting: Props | 0 | 0 | 8
  Sitting: Stable sit | 13 | 0 | 19
  Sitting: Pivots (rotates) | 63 | 0 | 15
  Ability to Kick: No kicking | 0 | 68 | 18
  Ability to Kick: Kick horizontally legs do not lift | 13 | 32 | 29
  Ability to Kick: Upward (vertically) | 0 | 0 | 10
  Ability to Kick: Touches leg | 0 | 0 | 11
  Ability to Kick: Touches toes | 88 | 0 | 32
  Rolling: No Rolling | 25 | 91 | 27
  Rolling: Rolling to Side | 0 | 9 | 37
  Rolling: Prone to Supine | 13 | 0 | 5
  Rolling: Supine to Prone | 63 | 0 | 31
  Crawling: Does not Lift Head | 63 | 100 | 81
  Crawling: On Elbow | 0 | 0 | 13
  Crawling: On Outstretched Hand | 0 | 0 | 2
  Crawling: Crawling Flat on Abdomen | 13 | 0 | 3
  Crawling: Crawling on Hands and Knees | 25 | 0 | 2
  Standing: Does not support weight | 38 | 100 | 79
  Standing: Supports weight | 13 | 0 | 11
  Standing: Stands with support | 25 | 0 | 10
  Standing: Stands unaided | 25 | 0 | 0
  Walking: No Walking | 75 | 100 | 95
  Walking: Bouncing | 0 | 0 | 0
  Walking: Cruising (Walks Holding on) | 13 | 0 | 5
  Walking: Walking Independently | 13 | 0 | 0
  Voluntary Grasp:No Grasp | 0 | 14 | 6
  Voluntary Grasp:Uses Whole Hand | 0 | 55 | 18
  Voluntary Grasp:Index Finger&Thumb;Immature Grasp | 0 | 14 | 21
  Voluntary Grasp:Pincer Grasp | 100 | 18 | 52

11. Secondary Outcome: Number of Participants Who Died or Met Permanent Ventilation
Description: Permanent ventilation was defined as tracheostomy or >=16 hours of ventilator support per day continuously for >21 days in the absence of an acute reversible event.
Time Frame: MMDR Period: Up to Day 1800
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Infantile SMA Onset CS3A | Infantile SMA Onset CS3B Previous Control | Infantile SMA Onset CS3B Previous ISIS 396443 | Later SMA Onset CS4 Previous Control | Later SMA Onset CS12 Type 2 | Later SMA Onset CS4 Previous ISIS 396443 | Later SMA Onset 232SM202 | Infantile SMA Onset 232SM202 | Later SMA Onset CS12 Type 3
Number analyzed (Participants) | 13 | 24 | 65 | 42 | 20 | 83 | 8 | 12 | 25
Participants | 0 | 6 | 11 | 1 | 0 | 1 | 0 | 2 | 0

12. Secondary Outcome: Number of Participants Not Requiring Permanent Ventilation
Description: as for outcome 11
Time Frame: MMDR Period: Up to Day 1800
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Infantile SMA Onset CS3A | Infantile SMA Onset CS3B Previous Control | Infantile SMA Onset CS3B Previous ISIS 396443 | Infantile SMA Onset 232SM202 | Later SMA Onset CS12 Type 2 | Later SMA Onset CS4 Previous Control | Later SMA Onset CS4 Previous ISIS 396443 | Later SMA Onset CS12 Type 3 | Later SMA Onset 232SM202
Number analyzed (Participants) | 13 | 24 | 65 | 12 | 20 | 42 | 83 | 25 | 8
Participants | 13 | 20 | 61 | 11 | 20 | 42 | 83 | 25 | 8

13. Secondary Outcome: Change From Baseline in Children's Hospital of Philadelphia Infant Test of Neuromuscular Disorders (CHOP INTEND) Motor Function Scale
Description: The CHOP INTEND test is designed to evaluate the motor skills of infants with significant motor weakness, including infants with SMA. Participants who are ≥2 years will be continued to be assessed until a CHOP INTEND maximum score of 64 is achieved. It includes 16 items structured to move from easiest to hardest with the grading including gravity eliminated (lower scores) to antigravity movements (higher scores). All item scores range from 0 (worst) to 4 (best). Total scores range from 0 to 64, with higher scores indicating better movement functioning.
Time Frame: Baseline, Day 2198
Population: The safety analysis set included all participants who were enrolled and received at least 1 dose of nusinersen or underwent sham procedure during CS11. 'Overall number of participants analyzed' signifies number of participants with data available for OM analysis. 'Number analyzed' signifies number of participants with data available for analysis at specified time point. Only CS3A and CS3B arm groups were planned to be analyzed for this OM.
Measure: Mean (Standard Deviation); unit: score on scale
Groups:
- Infantile SMA Onset CS3A: Participants who entered the study after receiving nusinersen in the open-label study ISIS 396443-CS3A received maintenance doses of nusinersen approximately every 4 months according to the MMDR dosing schedule.
- Infantile SMA Onset CS3B Previous Control: Participants who entered the study after receiving sham procedures in the double-blind study ISIS 396443-CS3B received 4 loading doses of nusinersen administered by IT injection on Days 1, 15, 29, and 64 (±1 day) followed by maintenance doses of nusinersen approximately every 4 months according to the MMDR dosing schedule.
- Infantile SMA Onset CS3B Previous ISIS 396443: Participants who entered the study after receiving nusinersen in the double-blind study ISIS 396443-CS3B received 3 sham procedures on Days 1, 15, and 64 and 1 loading dose of nusinersen administered by IT injection on Day 29 (±1 day) followed by maintenance doses of nusinersen approximately every 4 months according to the MMDR dosing schedule.
Arm/Group | Infantile SMA Onset CS3A | Infantile SMA Onset CS3B Previous Control | Infantile SMA Onset CS3B Previous ISIS 396443
Number analyzed (Participants) | 13 | 24 | 65
score on scale
  Baseline | 47.4 (13.09) | 17.3 (9.71) | 38.8 (9.43)
  Change at Day 2198: number analyzed (Participants) | 1 | 10 | 29
  Change at Day 2198 | -6.0 (NA) — Since only one participant was evaluable at Day 2198, the standard deviation (SD) could not be estimated. | 11.5 (12.21) | 4.7 (14.18)

14. Secondary Outcome: Change From Baseline in Hammersmith Functional Motor Scale Expanded (HFMSE) Total Score
Description: The HFMSE consists of 33 scored activities used to assess motor function in children with SMA. Participants were asked to do a specific activity (such as rolling) and they were then graded on the quality and execution of that movement on a scale of 0=being unable, 1=performed with some compensation, and 2=unaided. The overall score is the sum of the scores for all activities with a maximum achievable score of 66. Higher scores indicate increased motor function.
Time Frame: MMDR Period: Baseline, MMDR Day 1800
Population: The safety analysis set included all participants who were enrolled and received at least 1 dose of nusinersen or underwent sham procedure during CS11. 'Overall number of participants analyzed' signifies number of participants with data available for outcome measure analysis. 'Number analyzed' signifies number of participants with data available for analysis at specified timepoint.
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Infantile SMA Onset CS3A | Infantile SMA Onset CS3B Previous Control | Infantile SMA Onset CS3B Previous ISIS 396443 | Infantile SMA Onset 232SM202 | Later SMA Onset CS12 Type 2 | Later SMA Onset CS12 Type 3 | Later SMA Onset CS4 Previous Control | Later SMA Onset CS4 Previous ISIS 396443 | Later SMA Onset 232SM202
Number analyzed (Participants) | 13 | 17 | 49 | 12 | 20 | 23 | 42 | 81 | 8
score on scale
  Baseline | 14.5 (13.75) | 0.0 (0.0) | 7.3 (6.88) | 6.8 (6.06) | 25.6 (14.23) | 53.6 (8.24) | 21.1 (7.75) | 26.1 (10.99) | 24.5 (12.64)
  Change at MMDR Day 1800: number analyzed (Participants) | 10 | 9 | 31 | 8 | 12 | 17 | 19 | 45 | 6
  Change at MMDR Day 1800 | 3.4 (5.93) | 0.4 (0.88) | 6.0 (9.12) | -2.3 (3.37) | -7.0 (6.03) | -2.4 (3.41) | -4.7 (7.20) | -6.2 (6.36) | -1.2 (9.83)

15. Secondary Outcome: Change From Baseline in Revised Upper Limb Module (RULM) Total Score
Description: RULM Test is used in participants with SMA to assess upper limb functional ability items and has total of 20 items with an entry item that serves as functional class identification and does not contribute to total score. Remaining 19 scorable items reflect different functional domains and graded on 3-point system with score of 0 (unable), 1 (able, with modification), and 2 (able, no difficulty). There is only 1 item that is scored as a can/cannot score, with 1 as the highest score. Scorable items are summed for total score (0-37), higher scores indicating increased upper limb function. Positive change from baseline indicates improvement.
Time Frame: MMDR Period: Baseline, MMDR Day 1800
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Infantile SMA Onset CS3A | Infantile SMA Onset CS3B Previous Control | Infantile SMA Onset CS3B Previous ISIS 396443 | Infantile SMA Onset 232SM202 | Later SMA Onset CS12 Type 2 | Later SMA Onset CS12 Type 3 | Later SMA Onset CS4 Previous Control | Later SMA Onset CS4 Previous ISIS 396443 | Later SMA Onset 232SM202
Number analyzed (Participants) | 11 | 6 | 18 | 11 | 20 | 18 | 42 | 80 | 8
score on scale
  Baseline | 11.8 (7.24) | 1.7 (1.63) | 10.3 (6.05) | 7.6 (6.23) | 24.1 (6.14) | 35.9 (1.91) | 21.1 (4.26) | 23.9 (5.69) | 21.4 (8.60)
  Change at MMDR Day 1800: number analyzed (Participants) | 9 | 3 | 12 | 6 | 13 | 9 | 20 | 45 | 6
  Change at MMDR Day 1800 | 9.1 (4.70) | 0.7 (0.58) | 10.0 (5.38) | 3.3 (5.01) | 0.4 (3.23) | 0.9 (1.76) | 2.4 (3.97) | 1.2 (3.72) | 3.2 (2.71)

16. Secondary Outcome: Change From Baseline in Total Distance Walked Over Time as Assessed by 6-Minute Walk Test (6MWT)
Description: The 6MWT measures the distance an individual can walk over a total of six minutes on a hard, flat surface. The goal is for the individual to walk as far as possible in six minutes.
Time Frame: Baseline, Day 2670
Population: The safety analysis set included all participants who were enrolled and received at least 1 dose of nusinersen or underwent sham procedure during CS11. 'Overall number of participants analyzed' signifies number of participants with data available for outcome measure analysis. 'Number analyzed' signifies number of participants with data available for analysis at specified timepoint. Only CS12 Type 2 and CS12 Type 3 arm groups were planned to be analysed for this end point.
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Later SMA Onset CS12 Type 2 | Later SMA Onset CS12 Type 3
Number analyzed (Participants) | 1 | 13
meters
  Baseline | 0 (NA) — Due to 1 evaluable participant, SD was not estimated | 253.3 (182.74)
  Change at Day 2670: number analyzed (Participants) | 1 | 6
  Change at Day 2670 | 156.5 (NA) — Due to 1 evaluable participant, SD was not estimated | 91.5 (49.07)

17. Secondary Outcome: Number of Participants Who Experienced Contracture Assesment
Description: Contracture assessment is performed to assess the motor performance in SMA. The number of participants who experienced at least one contracture at any location and severe contractures in any of the five locations (hip flexors, knee flexors, ankle planter flexors, elbow flexors, forearm flexors) are reported in this outcome measure.
Time Frame: MMDR Period: At MMDR Day 1800
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Infantile SMA Onset CS3A | Infantile SMA Onset CS3B Previous Control | Infantile SMA Onset CS3B Previous ISIS 396443 | Infantile SMA Onset 232SM202 | Later SMA Onset CS12 Type 2 | Later SMA Onset CS12 Type 3 | Later SMA Onset CS4 Previous Control | Later SMA Onset CS4 Previous ISIS 396443 | Later SMA Onset 232SM202
Number analyzed (Participants) | 10 | 10 | 41 | 8 | 13 | 18 | 20 | 45 | 5
Participants
  At least one contracture at any location | 9 | 10 | 36 | 8 | 13 | 8 | 19 | 44 | 5
  Severe contractures in any of the five locations | 3 | 3 | 16 | 4 | 6 | 1 | 9 | 16 | 2

18. Secondary Outcome: Change From Baseline in Compound Muscular Action Potential (CMAP)
Description: CMAP is an electrophysiological technique that can be used to determine the approximate number of motor neurons in a muscle or group of muscles. Peroneal amplitude (PA) and ulnar amplitude (UA) data is reported in this OM. Score <0 indicated worse response and >0 indicated better response than the normal matched population. Score change <0 indicated worsening and >0 indicated improvement as compared to baseline.
Time Frame: MMDR Period: Baseline, MMDR Day 1800
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: millivolt (mV)
Arm/Group | Infantile SMA Onset CS3A | Infantile SMA Onset CS3B Previous Control | Infantile SMA Onset CS3B Previous ISIS 396443 | Infantile SMA Onset 232SM202 | Later SMA Onset CS12 Type 2 | Later SMA Onset CS12 Type 3 | Later SMA Onset CS4 Previous Control | Later SMA Onset CS4 Previous ISIS 396443 | Later SMA Onset 232SM202
Number analyzed (Participants) | 13 | 22 | 60 | 8 | 20 | 23 | 33 | 62 | 6
millivolt (mV)
  PA: Baseline: number analyzed (Participants) | 13 | 22 | 60 | 8 | 19 | 22 | 33 | 62 | 6
  PA: Baseline | 3.02 (2.207) | 0.35 (0.517) | 1.91 (1.367) | 0.94 (0.929) | 1.89 (1.369) | 2.71 (1.318) | 2.00 (2.189) | 1.97 (1.586) | 1.35 (0.948)
  PA: Change at MMDR Day 1800: number analyzed (Participants) | 9 | 5 | 34 | 6 | 7 | 13 | 13 | 28 | 2
  PA: Change at MMDR Day 1800 | -0.41 (1.290) | 0.10 (0.243) | 0.30 (1.395) | 0.92 (1.901) | -0.59 (1.069) | -0.08 (1.799) | 0.22 (4.832) | -0.28 (0.924) | 0.10 (1.414)
  UA: Baseline | 1.52 (1.563) | 0.20 (0.205) | 0.85 (0.944) | 0.99 (0.861) | 2.81 (1.723) | 6.76 (2.448) | 1.69 (1.133) | 2.71 (2.161) | 1.25 (0.935)
  UA: Change at MMDR Day 1800: number analyzed (Participants) | 9 | 5 | 35 | 6 | 7 | 14 | 13 | 28 | 2
  UA: Change at MMDR Day 1800 | 0.45 (0.837) | 0.20 (0.188) | 0.67 (1.261) | 0.15 (0.436) | 0.04 (0.957) | 0.04 (1.641) | 0.32 (1.127) | 0.52 (1.600) | 2.77 (2.729)

19. Secondary Outcome: Change From Baseline in Body Length
Description: Participants were analyzed for change in growth parameter of body length to evaluate clinical efficacy. The body length was calculated using either WHO or Centers for Disease Control and Prevention (CDC) scales. The CDC scale allows to calculate the body length up to 20 years, while the WHO scale allows to calculate it only up to 10 years.
Time Frame: MMDR Period: up to Day 1800
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: centimeters (cm)
Arm/Group | Infantile SMA Onset CS3A | Infantile SMA Onset CS3B Previous Control | Infantile SMA Onset CS3B Previous ISIS 396443 | Infantile SMA Onset 232SM202 | Later SMA Onset CS12 Type 2 | Later SMA Onset CS12 Type 3 | Later SMA Onset CS4 Previous Control | Later SMA Onset CS4 Previous ISIS 396443 | Later SMA Onset 232SM202
Number analyzed (Participants) | 4 | 7 | 14 | 6 | 4 | 1 | 8 | 23 | 2
centimeters (cm) | 24.2 (2.86) | 19.9 (6.99) | 29.4 (6.38) | 18.8 (10.92) | 18.8 (8.54) | 23.1 (0) | 23.7 (7.06) | 24.6 (10.60) | -10.3 (57.63)

20. Secondary Outcome: Change From Baseline in Weight
Description: Participants were analyzed for change in growth parameter of weight to evaluate clinical efficacy. The weight was calculated using either WHO or CDC scales. The CDC scale allows to calculate the weight up to 20 years, while the WHO scale allows to calculate it only up to 10 years.
Time Frame: MMDR Period: up to Day 1800
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: kilograms (kg)
Groups:
- Infantile SMA Onset CS3A: Participants who received nusinersen in study ISIS 396443-CS3A, in an open-label period, received maintenance doses of nusinersen, intrathecal (IT) injection, on days 1, 120, 240, 360, 480, 600, 720, 840, 960, 1080, 1200, 1320, 1440, 1560, and 1680 in MMDR period of this study.
Arm/Group | Infantile SMA Onset CS3A | Infantile SMA Onset CS3B Previous Control | Infantile SMA Onset CS3B Previous ISIS 396443 | Infantile SMA Onset 232SM202 | Later SMA Onset CS12 Type 2 | Later SMA Onset CS12 Type 3 | Later SMA Onset CS4 Previous Control | Later SMA Onset CS4 Previous ISIS 396443 | Later SMA Onset 232SM202
Number analyzed (Participants) | 9 | 11 | 43 | 8 | 13 | 20 | 20 | 50 | 6
kilograms (kg) | 9.8 (3.48) | 7.7 (4.39) | 9.3 (3.25) | 9.5 (7.04) | 15.1 (5.96) | 13.8 (14.88) | 15.4 (8.05) | 15.2 (7.38) | 11.7 (8.09)

21. Secondary Outcome: Change From Baseline in Weight for Age Percentile
Description: Participants who were below the age of 36 months were analyzed for change in growth parameter of weight for age to evaluate clinical efficacy. The weight for age percentile was calculated using either WHO or CDC scales. The CDC scale allows to calculate the weight for age percentile up to 20 years, while the WHO scale allows to calculate it only up to 10 years.
Time Frame: MMDR Period: up to Day 1800
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: percentile
Arm/Group | Infantile SMA Onset CS3A | Infantile SMA Onset CS3B Previous Control | Infantile SMA Onset CS3B Previous ISIS 396443 | Infantile SMA Onset 232SM202 | Later SMA Onset CS12 Type 2 | Later SMA Onset CS12 Type 3 | Later SMA Onset CS4 Previous Control | Later SMA Onset CS4 Previous ISIS 396443 | Later SMA Onset 232SM202
Number analyzed (Participants) | 8 | 11 | 43 | 6 | 0 | 0 | 9 | 14 | 6
percentile | 5.7 (27.30) | -5.3 (28.97) | 0.3 (28.55) | -0.7 (25.32) |  |  | 0.9 (17.22) | 20.2 (28.15) | 4.0 (33.11)

22. Secondary Outcome: Percentage of CMAP Responders
Description: CMAP is an electrophysiological technique that can be used to determine the approximate number of motor neurons in a muscle or group of muscles. A participant was defined as a responder if they had a peroneal amplitude ≥1 mV at last visit (including the amplitude ≥1 mV at baseline and also demonstrated as such at last visit).
Time Frame: MMDR Period: At Day 1800
Population: as for outcome 9
Measure: Number; unit: percentage of responders
Arm/Group | Infantile SMA Onset CS3A | Infantile SMA Onset CS3B Previous Control | Infantile SMA Onset CS3B Previous ISIS 396443 | Infantile SMA Onset 232SM202 | Later SMA Onset CS12 Type 2 | Later SMA Onset CS12 Type 3 | Later SMA Onset CS4 Previous Control | Later SMA Onset CS4 Previous ISIS 396443 | Later SMA Onset 232SM202
Number analyzed (Participants) | 13 | 22 | 60 | 12 | 20 | 24 | 42 | 81 | 8
percentage of responders | 85 | 0 | 72 | 33 | 65 | 67 | 60 | 51 | 25

23. Secondary Outcome: Number of Participants Who Achieved Motor Milestones
Description: Motor milestones were measured based on WHO criteria. The WHO motor milestones are a set of six milestones in motor development, all of which would be expected to be attained by 24 months of age in healthy children. The individual milestones are: sitting without support (SWS), standing with assistance (SWA), hands and knees crawling (HKC), and walking alone (WA).
Time Frame: MMDR Period: up to Day 1800
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Infantile SMA Onset CS3A | Infantile SMA Onset CS3B Previous Control | Infantile SMA Onset CS3B Previous ISIS 396443 | Infantile SMA Onset 232SM202 | Later SMA Onset CS12 Type 2 | Later SMA Onset CS12 Type 3 | Later SMA Onset CS4 Previous Control | Later SMA Onset CS4 Previous ISIS 396443 | Later SMA Onset 232SM202
Number analyzed (Participants) | 12 | 22 | 60 | 12 | 20 | 24 | 42 | 81 | 8
Participants
  SWS:Achieved at Baseline&Maintained to Last Visit | 5 | 0 | 16 | 3 | 13 | 23 | 27 | 58 | 5
  SWS:Inability at Baseline, Achieved at Last visit | 3 | 0 | 11 | 0 | 0 | 0 | 0 | 0 | 0
  HKC:Achieved at Baseline&Maintained to Last Visit | 1 | 0 | 0 | 0 | 4 | 20 | 3 | 18 | 2
  HKC: Inability at Baseline, Achieved at Last Visit | 0 | 0 | 4 | 0 | 0 | 1 | 1 | 2 | 1
  SWA:Achieved at Baseline&Maintained to Last Visit | 1 | 0 | 3 | 0 | 1 | 20 | 3 | 3 | 1
  SWA:Inability at Baseline, Achieved at Last Visit | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0
  WA: Achieved at Baseline&Maintained to Last Visit | 1 | 0 | 0 | 0 | 1 | 16 | 1 | 2 | 1
  WA: Inability at Baseline, Achieved at Last Visit | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0

24. Secondary Outcome: Number of Participants Who Achieved Standing Alone and Walking With Assistance
Description: Motor milestones were measured based on WHO criteria. The WHO motor milestones are a set of six milestones in motor development, all of which would be expected to be attained by 24 months of age in healthy children. The individual milestones are: SWS, SWA, HKC, WWA, WA and standing alone (SA). SA and WWA were assessed in this outcome measure.
Time Frame: MMDR Period: up to Day 1800
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Infantile SMA Onset CS3A | Infantile SMA Onset CS3B Previous Control | Infantile SMA Onset CS3B Previous ISIS 396443 | Infantile SMA Onset 232SM202 | Later SMA Onset CS12 Type 2 | Later SMA Onset CS12 Type 3 | Later SMA Onset CS4 Previous Control | Later SMA Onset CS4 Previous ISIS 396443 | Later SMA Onset 232SM202
Number analyzed (Participants) | 12 | 22 | 60 | 12 | 20 | 24 | 42 | 81 | 8
Participants
  SA: Achieved at Baseline & Maintained to Last Visit | 1 | 0 | 0 | 0 | 1 | 19 | 1 | 2 | 1
  SA: Inability at Baseline, Achieved at Last Visit | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
  WWA: Achieved at Baseline & Maintained to Last Visit | 1 | 0 | 1 | 0 | 1 | 19 | 2 | 2 | 1
  WWA: Inability at Baseline, Achieved at Last Visit | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0

25. Secondary Outcome: Total Number of Hospitalizations Due to Serious Respiratory Events
Description: Total number of hospitalizations is total number of serious events that occurred during study for all participants under each group. For a participant with multiple SAEs which started at the same date and led to hospitalization, it is counted as one hospitalization.
Time Frame: Up to day 2520
Population: as for outcome 14
Measure: Number; unit: number of hospitalizations
Arm/Group | Infantile SMA Onset CS3A | Infantile SMA Onset CS3B Previous Control | Infantile SMA Onset CS3B Previous ISIS 396443 | Infantile SMA Onset 232SM202 | Later SMA Onset CS12 Type 2 | Later SMA Onset CS12 Type 3 | Later SMA Onset CS4 Previous Control | Later SMA Onset CS4 Previous ISIS 396443 | Later SMA Onset 232SM202
Number analyzed (Participants) | 13 | 24 | 65 | 12 | 20 | 25 | 42 | 83 | 8
number of hospitalizations
  Day 1-360 | 2 | 12 | 30 | 2 | 0 | 0 | 2 | 0 | 0
  Day 361-720: number analyzed (Participants) | 13 | 22 | 61 | 12 | 20 | 25 | 42 | 83 | 8
  Day 361-720 | 2 | 13 | 18 | 1 | 1 | 0 | 2 | 1 | 0
  Day 721-1080: number analyzed (Participants) | 12 | 22 | 60 | 12 | 19 | 24 | 42 | 81 | 8
  Day 721-1080 | 0 | 15 | 12 | 0 | 0 | 0 | 1 | 2 | 0
  Day 1081-1440: number analyzed (Participants) | 12 | 21 | 59 | 11 | 18 | 23 | 39 | 78 | 8
  Day 1081-1440 | 1 | 0 | 4 | 1 | 1 | 0 | 1 | 1 | 0
  Day 1441-1800: number analyzed (Participants) | 12 | 18 | 55 | 10 | 18 | 23 | 38 | 76 | 7
  Day 1441-1800 | 2 | 2 | 2 | 2 | 0 | 0 | 0 | 3 | 0
  Day 1801-2160: number analyzed (Participants) | 12 | 16 | 52 | 6 | 18 | 23 | 32 | 71 | 1
  Day 1801-2160 | 1 | 1 | 7 | 0 | 0 | 0 | 0 | 1 | 0
  Day 2161-2520: number analyzed (Participants) | 13 | 10 | 39 | 0 | 12 | 20 | 18 | 48 | 0
  Day 2161-2520 | 0 | 0 | 1 |  | 0 | 0 | 0 | 0 |

26. Secondary Outcome: Total Number of Hospitalizations Due to Serious Adverse Events
Description: as for outcome 25
Time Frame: Up to day 2520
Population: as for outcome 14
Measure: Number; unit: number of hospitalizations
Arm/Group | Infantile SMA Onset CS3A | Infantile SMA Onset CS3B Previous Control | Infantile SMA Onset CS3B Previous ISIS 396443 | Infantile SMA Onset 232SM202 | Later SMA Onset CS12 Type 2 | Later SMA Onset CS12 Type 3 | Later SMA Onset CS4 Previous Control | Later SMA Onset CS4 Previous ISIS 396443 | Later SMA Onset 232SM202
Number analyzed (Participants) | 13 | 24 | 65 | 12 | 20 | 25 | 42 | 83 | 8
number of hospitalizations
  Day 1-360 | 6 | 26 | 89 | 12 | 2 | 0 | 10 | 8 | 3
  Day 361-720: number analyzed (Participants) | 13 | 22 | 61 | 12 | 20 | 25 | 42 | 83 | 8
  Day 361-720 | 6 | 19 | 64 | 4 | 7 | 2 | 10 | 12 | 2
  Day 721-1080: number analyzed (Participants) | 12 | 22 | 60 | 12 | 19 | 24 | 42 | 81 | 8
  Day 721-1080 | 5 | 29 | 63 | 7 | 2 | 0 | 21 | 21 | 1
  Day 1081-1440: number analyzed (Participants) | 12 | 21 | 59 | 11 | 18 | 23 | 39 | 78 | 8
  Day 1081-1440 | 2 | 10 | 36 | 4 | 5 | 1 | 6 | 10 | 3
  Day 1441-1800: number analyzed (Participants) | 12 | 18 | 55 | 10 | 18 | 23 | 38 | 76 | 7
  Day 1441-1800 | 4 | 10 | 19 | 3 | 3 | 0 | 5 | 18 | 0
  Day 1801-2160: number analyzed (Participants) | 12 | 16 | 52 | 6 | 18 | 23 | 32 | 71 | 1
  Day 1801-2160 | 1 | 8 | 32 | 0 | 2 | 2 | 6 | 13 | 0
  Day 2161-2520: number analyzed (Participants) | 13 | 10 | 39 | 0 | 12 | 20 | 18 | 48 | 0
  Day 2161-2520 | 0 | 1 | 14 |  | 0 | 0 | 1 | 2 |

27. Secondary Outcome: Percent of Time in Hospitalization
Time Frame: Upto day 2160
Population: as for outcome 14
Measure: Median (Full Range); unit: percentage of days
Arm/Group | Infantile SMA Onset CS3A | Infantile SMA Onset CS3B Previous Control | Infantile SMA Onset CS3B Previous ISIS 396443 | Infantile SMA Onset 232SM202 | Later SMA Onset CS12 Type 2 | Later SMA Onset CS12 Type 3 | Later SMA Onset CS4 Previous Control | Later SMA Onset CS4 Previous ISIS 396443 | Later SMA Onset 232SM202
Number analyzed (Participants) | 13 | 22 | 60 | 12 | 20 | 24 | 42 | 81 | 8
percentage of days
  Day 1-360 | 0.00 [0.00 to 2.0] | 1.11 [0.00 to 16.7] | 0.28 [0.00 to 22.8] | 0.28 [0.00 to 11.4] | 0.00 [0.00 to 2.5] | 0.00 [0.00 to 0.8] | 0.00 [0.00 to 4.4] | 0.00 [0.00 to 6.4] | 0.0 [0.0 to 2.8]
  Day 361-720: number analyzed (Participants) | 12 | 22 | 60 | 12 | 18 | 24 | 42 | 80 | 8
  Day 361-720 | 0.28 [0.00 to 4.7] | 2.08 [0.00 to 17.2] | 0.56 [0.00 to 19.2] | 0.00 [0.00 to 7.8] | 0.00 [0.00 to 3.1] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 10.3] | 0.00 [0.00 to 29.7] | 0.0 [0.0 to 2.5]
  Day 721-1080: number analyzed (Participants) | 12 | 20 | 59 | 12 | 18 | 23 | 39 | 78 | 8
  Day 721-1080 | 0.00 [0.00 to 1.7] | 0.00 [0.00 to 7.5] | 0.00 [0.00 to 31.3] | 0.00 [0.00 to 20.3] | 0.00 [0.00 to 6.1] | 0.00 [0.00 to 1.4] | 0.00 [0.00 to 3.6] | 0.00 [0.00 to 12.2] | 0.0 [0.0 to 11.4]
  Day 1081-1440: number analyzed (Participants) | 12 | 17 | 54 | 11 | 18 | 23 | 36 | 75 | 8
  Day 1081-1440 | 0.00 [0.00 to 0.8] | 0.00 [0.00 to 7.5] | 0.00 [0.00 to 9.7] | 0.00 [0.00 to 48.6] | 0.00 [0.00 to 1.9] | 0.00 [0.00 to 0.8] | 0.00 [0.00 to 5.8] | 0.00 [0.00 to 35.3] | 0.69 [0.0 to 1.9]
  Day 1441-1800: number analyzed (Participants) | 12 | 15 | 50 | 10 | 17 | 23 | 33 | 70 | 7
  Day 1441-1800 | 0.00 [0.00 to 8.3] | 0.00 [0.00 to 20.2] | 0.00 [0.00 to 22.6] | 0.00 [0.00 to 12.1] | 0.00 [0.00 to 2.0] | 0.00 [0.00 to 0.8] | 0.00 [0.00 to 5.3] | 0.00 [0.00 to 8.9] | 0.00 [0.00 to 1.7]
  Day 1801-2160: number analyzed (Participants) | 7 | 8 | 19 | 6 | 10 | 18 | 9 | 31 | 1
  Day 1801-2160 | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00]

28. Secondary Outcome: Change From Baseline in Cobb-Angle on X-Ray of the Thoracolumbar Spine by Visit
Description: Cobb angle is a measurement of the degree of side-to-side spinal curvature used to define scoliosis.
Time Frame: MMDR Period: Baseline, MMDR Day 1800
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: degree
Arm/Group | Infantile SMA Onset CS3A | Infantile SMA Onset CS3B Previous Control | Infantile SMA Onset CS3B Previous ISIS 396443 | Infantile SMA Onset 232SM202 | Later SMA Onset CS12 Type 2 | Later SMA Onset CS12 Type 3 | Later SMA Onset CS4 Previous Control | Later SMA Onset CS4 Previous ISIS 396443 | Later SMA Onset 232SM202
Number analyzed (Participants) | 8 | 11 | 42 | 8 | 12 | 10 | 35 | 67 | 5
degree
  Baseline | 22.7 (17.86) | 16.6 (13.38) | 34.8 (18.43) | 49.2 (13.19) | 38.5 (27.36) | 29.8 (25.09) | 24.3 (19.08) | 26.8 (20.33) | 33.0 (16.94)
  Change at MMDR day 1800: number analyzed (Participants) | 4 | 4 | 26 | 5 | 4 | 7 | 15 | 30 | 1
  Change at MMDR day 1800 | 29.8 (9.46) | 16.9 (27.27) | 13.0 (29.91) | -11.6 (24.65) | -3.8 (17.01) | 4.0 (7.78) | 19.8 (30.83) | 18.8 (30.30) | -13.8 (0)

29. Secondary Outcome: Pediatric Quality of Life Inventory (PedsQL) Questionnaires Total Score by Domain
Description: Items on the PedsQL generic core scale are reverse scored and transformed to a 0-100 scale. The PedsQL parent (P) and self (S) reported questionnaire was collected for participants from 2 to 25 years of age. Four dimensions were collected: Physical, Emotional, Social and School functioning and each item was scored on a 5 point ordinal scale. 0 (never) =100, 1 (almost never) = 75, 2 (sometimes)= 50, 3 (often) = 25, 4 (almost always) = 0. A total score was calculated as the sum of all the items over the number of items answered on all the scales. If more than 50% of items or more were missing, the scale score was not computed. Higher scores indicated better health related quality of life.
Time Frame: MMDR Period: At Day 1800
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Infantile SMA Onset CS3A | Infantile SMA Onset CS3B Previous Control | Infantile SMA Onset CS3B Previous ISIS 396443 | Infantile SMA Onset 232SM202 | Later SMA Onset CS12 Type 2 | Later SMA Onset CS12 Type 3 | Later SMA Onset CS4 Previous Control | Later SMA Onset CS4 Previous ISIS 396443 | Later SMA Onset 232SM202
Number analyzed (Participants) | 8 | 11 | 42 | 7 | 8 | 11 | 20 | 50 | 6
score on scale
  S: Physical Functioning Report: number analyzed (Participants) | 8 | 6 | 28 | 7 | 8 | 11 | 20 | 50 | 5
  S: Physical Functioning Report | 37.1 (11.26) | 22.4 (31.52) | 47.5 (25.31) | 32.6 (20.48) | 37.5 (13.68) | 52.7 (16.94) | 45.4 (13.85) | 39.7 (17.97) | 53.7 (24.46)
  S: Emotional Functioning Report: number analyzed (Participants) | 8 | 6 | 29 | 7 | 8 | 11 | 20 | 50 | 5
  S: Emotional Functioning Report | 61.9 (12.52) | 61.7 (26.39) | 63.3 (20.71) | 67.1 (19.55) | 79.2 (14.41) | 78.0 (21.24) | 84.6 (15.42) | 74.5 (22.80) | 67.0 (16.43)
  S: Social Functioning: number analyzed (Participants) | 8 | 6 | 28 | 7 | 8 | 11 | 20 | 50 | 5
  S: Social Functioning | 67.5 (22.83) | 50.8 (41.52) | 67.1 (22.87) | 75.7 (20.09) | 77.7 (11.66) | 80.8 (13.11) | 83.3 (15.07) | 76.3 (13.88) | 80.0 (12.25)
  S: School/Work Functioning Report: number analyzed (Participants) | 8 | 6 | 28 | 5 | 8 | 11 | 20 | 50 | 5
  S: School/Work Functioning Report | 54.4 (14.25) | 40.8 (33.23) | 66.1 (17.66) | 71.4 (14.64) | 77.3 (13.33) | 77.8 (15.09) | 81.8 (14.89) | 77.1 (15.22) | 82.0 (11.51)
  P: Physical Functioning Report: number analyzed (Participants) | 8 | 10 | 42 | 7 | 8 | 9 | 20 | 49 | 6
  P: Physical Functioning Report | 25.0 (27.55) | 19.1 (24.54) | 24.9 (22.77) | 32.6 (30.07) | 28.6 (14.31) | 46.1 (21.47) | 35.2 (18.19) | 33.5 (18.41) | 20.8 (5.82)
  P: Emotional Functioning Report: number analyzed (Participants) | 8 | 10 | 42 | 7 | 8 | 9 | 20 | 49 | 6
  P: Emotional Functioning Report | 68.1 (13.08) | 69.5 (17.23) | 58.7 (14.90) | 65.0 (26.46) | 72.7 (19.75) | 71.8 (19.84) | 78.0 (18.74) | 78.2 (19.60) | 74.2 (11.14)
  P: Social Functioning Report: number analyzed (Participants) | 8 | 10 | 42 | 7 | 8 | 9 | 20 | 49 | 6
  P: Social Functioning Report | 47.5 (12.82) | 54.0 (23.66) | 51.3 (20.06) | 64.3 (22.63) | 71.9 (24.46) | 72.1 (16.96) | 70.0 (20.65) | 71.0 (17.50) | 60.8 (13.20)
  P: School/Work Functioning Report: number analyzed (Participants) | 8 | 11 | 42 | 7 | 8 | 9 | 20 | 49 | 5
  P: School/Work Functioning Report | 48.8 (12.17) | 48.5 (31.23) | 51.4 (21.36) | 63.6 (18.64) | 76.5 (13.45) | 78.5 (18.44) | 78.8 (20.19) | 78.0 (14.75) | 79.2 (9.70)

30. Secondary Outcome: Change From Baseline in Assessment of Caregiver Experience With Neuromuscular Disease (ACEND) Questionnaire Total Score
Description: The ACEND is a questionnaire that includes a total of seven domains assessing physical impact (including feeding/grooming/dressing, sitting/play, transfers, and mobility) and general caregiver impact (including time, emotion, and finance) and each domain comprises several items. The total score (TS) for each domain will be calculated on a scale of 0 to 100. Higher scores indicate a greater impact on the caregiver.
Time Frame: MMDR Period: up to Day 1800
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Infantile SMA Onset CS3A | Infantile SMA Onset CS3B Previous Control | Infantile SMA Onset CS3B Previous ISIS 396443 | Infantile SMA Onset 232SM202 | Later SMA Onset CS12 Type 2 | Later SMA Onset CS12 Type 3 | Later SMA Onset CS4 Previous Control | Later SMA Onset CS4 Previous ISIS 396443 | Later SMA Onset 232SM202
Number analyzed (Participants) | 10 | 11 | 38 | 8 | 8 | 9 | 18 | 47 | 6
score on scale
  Feeding/Grooming/Dressing TS: Change MMDR Day1800 | 14.2 (21.56) | 0.6 (2.01) | 18.5 (22.07) | 9.2 (15.91) | 2.1 (14.82) | 0.6 (2.43) | 4.6 (18.90) | 5.9 (12.07) | 2.8 (7.72)
  Sitting/Play TS: Change at MMDR Day 1800 | 0.8 (10.29) | -0.4 (14.91) | 5.5 (28.01) | 1.5 (22.21) | 2.8 (12.04) | 0.0 (0.00) | -1.8 (16.48) | 1.7 (16.08) | -2.0 (4.90)
  Transfers TS: Change at MMDR Day 1800 | 0.4 (7.24) | 0.7 (1.62) | 0.0 (12.32) | -5.5 (6.68) | -5.8 (15.14) | 1.4 (9.48) | -3.6 (16.17) | 1.2 (18.16) | -4.0 (11.03)
  Mobility TS: Change at MMDR Day 1800 | -2.3 (14.93) | 0.5 (1.72) | 7.5 (22.52) | -12.1 (18.69) | -13.0 (13.83) | -2.2 (7.86) | 1.9 (18.47) | -5.8 (17.50) | 6.7 (20.66)
  Time TS: Change at MMDR Day 1800 | 4.4 (19.78) | 6.8 (24.76) | -0.7 (22.60) | -6.3 (21.65) | -2.4 (18.14) | 2.6 (18.36) | 1.4 (17.22) | 0.5 (16.78) | -6.3 (14.25)
  Emotion TS: Change at MMDR Day 1800 | 5.0 (14.80) | 6.3 (15.82) | -2.1 (20.98) | 2.1 (14.22) | -2.4 (21.00) | 1.0 (13.25) | 4.7 (12.73) | -2.5 (12.70) | -18.1 (12.01)
  Finance TS: Change at MMDR Day 1800 | -1.0 (17.29) | 7.3 (20.66) | -4.1 (22.17) | 4.4 (18.98) | -0.8 (20.70) | 4.1 (14.92) | 7.2 (17.92) | 2.1 (19.94) | -3.3 (8.16)

31. Secondary Outcome: Number of Participants With Disease-related Hospitalizations and AEs
Time Frame: MMDR Period: up to Day 1800
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Infantile SMA Onset CS3A | Infantile SMA Onset CS3B Previous Control | Infantile SMA Onset CS3B Previous ISIS 396443 | Infantile SMA Onset 232SM202 | Later SMA Onset CS12 Type 2 | Later SMA Onset CS12 Type 3 | Later SMA Onset CS4 Previous Control | Later SMA Onset CS4 Previous ISIS 396443 | Later SMA Onset 232SM202
Number analyzed (Participants) | 13 | 24 | 65 | 12 | 20 | 25 | 42 | 83 | 8
Participants
  Disease-related hospitalization | 6 | 9 | 27 | 5 | 9 | 0 | 13 | 23 | 3
  Disease-related AEs | 11 | 21 | 60 | 7 | 16 | 12 | 36 | 68 | 8

32. Secondary Outcome: Survival Rate
Description: Survival rate was defined as the percentage of participants alive during the study and was estimated from the Kaplan Meier (KM) curve for time to death.
Time Frame: MMDR Period: up to Day 1800
Population: All dosed population included all participants who received a dose of nusinersen or were in the sham treatment group. 'Overall number of participants analyzed' signifies number of participants with data available for outcome measure analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Infantile SMA Onset CS3A | Infantile SMA Onset CS3B Previous Control | Infantile SMA Onset CS3B Previous ISIS 396443 | Later SMA Onset CS4 Previous Control | Later SMA Onset CS4 Previous ISIS 396443 | Later SMA Onset 232SM202 | Later SMA Onset CS12 Type 2 | Infantile SMA Onset 232SM202 | Later SMA Onset CS12 Type 3
Number analyzed (Participants) | 13 | 24 | 65 | 42 | 83 | 8 | 20 | 12 | 25
percentage of participants | 100 | 79.16 | 87.69 | 97.61 | 98.79 | 100 | 100 | 91.66 | 100

ADVERSE EVENTS:
Time Frame: From Day 1 up to the end of the study (up to 2848 days)
Description: Safety analysis set included all participants who were enrolled and received at least 1 dose of nusinersen or underwent sham procedure during CS11.
Arm/Group | Infantile SMA Onset CS3A | Infantile SMA Onset CS3B Previous Control | Infantile SMA Onset CS3B Previous ISIS 396443 | Infantile SMA Onset 232SM202 | Later SMA Onset 232SM202 | Later SMA Onset CS12 Type 2 | Later SMA Onset CS12 Type 3 | Later SMA Onset CS4 Previous Control | Later SMA Onset CS4 Previous ISIS 396443
All-Cause Mortality (participants affected / at risk) | 0/13 | 5/24 | 8/65 | 1/12 | 0/8 | 0/20 | 0/25 | 1/42 | 1/83
Serious Adverse Events (participants affected / at risk) | 11/13 | 23/24 | 59/65 | 9/12 | 5/8 | 12/20 | 6/25 | 26/42 | 47/83
Other Adverse Events (participants affected / at risk) | 13/13 | 23/24 | 65/65 | 12/12 | 8/8 | 20/20 | 25/25 | 40/42 | 79/83
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Infantile SMA Onset CS3A (N=13) | Infantile SMA Onset CS3B Previous Control (N=24) | Infantile SMA Onset CS3B Previous ISIS 396443 (N=65) | Infantile SMA Onset 232SM202 (N=12) | Later SMA Onset 232SM202 (N=8) | Later SMA Onset CS12 Type 2 (N=20) | Later SMA Onset CS12 Type 3 (N=25) | Later SMA Onset CS4 Previous Control (N=42) | Later SMA Onset CS4 Previous ISIS 396443 (N=83)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Cardio-respiratory arrest (Cardiac disorders) | 0 | 2 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Supraventricular extrasystoles (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Wolff-parkinson-white syndrome (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cryptorchism (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Developmental hip dysplasia (Congenital, familial and genetic disorders) | 1 | 0 | 2 | 0 | 1 | 0 | 0 | 1 | 2
Laryngeal cleft (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Spinal muscular atrophy (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Talipes (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acetonaemic vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Colitis ulcerative (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0
Cyclic vomiting syndrome (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dental caries (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Faecaloma (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Gastritis haemorrhagic (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Gingival hypertrophy (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hiatus hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ileus (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Subileus (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 5 | 0 | 0 | 0 | 0 | 0 | 0
Complication associated with device (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Complication of device insertion (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Death (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Discomfort (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Generalised oedema (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Impaired healing (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Medical device discomfort (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 2 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Sudden death (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Anaphylactic reaction (Immune system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cytokine storm (Immune system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Acute sinusitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Adenovirus infection (Infections and infestations) | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Appendicitis perforated (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Bacterial infection (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Bronchiolitis (Infections and infestations) | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 4 | 0 | 0 | 0 | 0 | 1 | 2
Bronchitis pneumococcal (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cellulitis staphylococcal (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Clostridium difficile infection (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Coronavirus infection (Infections and infestations) | 0 | 1 | 3 | 0 | 0 | 0 | 0 | 1 | 0
Coronavirus pneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Covid-19 (Infections and infestations) | 0 | 0 | 3 | 1 | 0 | 0 | 0 | 0 | 1
Covid-19 pneumonia (Infections and infestations) | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Device related infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Enterovirus infection (Infections and infestations) | 0 | 1 | 6 | 1 | 0 | 0 | 0 | 3 | 0
Escherichia infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gastritis viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 4 | 0 | 0 | 0 | 0 | 2 | 1
Gastroenteritis adenovirus (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 2 | 1
Haemophilus infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Human bocavirus infection (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Incision site abscess (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 1 | 3
Intestinal sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Laryngitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 2 | 7 | 1 | 0 | 0 | 0 | 0 | 1
Lower respiratory tract infection viral (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Medical device site abscess (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Metapneumovirus infection (Infections and infestations) | 1 | 2 | 4 | 1 | 0 | 0 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Osteomyelitis chronic (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Otitis media (Infections and infestations) | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Otitis media acute (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Otitis media chronic (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Parainfluenzae virus infection (Infections and infestations) | 0 | 1 | 6 | 1 | 0 | 0 | 0 | 0 | 0
Periorbital cellulitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Peritonitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pharyngitis streptococcal (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pharyngotonsillitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumococcal bacteraemia (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 3 | 8 | 27 | 5 | 1 | 2 | 0 | 8 | 6
Pneumonia aspiration (Infections and infestations) | 0 | 2 | 6 | 0 | 0 | 0 | 0 | 1 | 0
Pneumonia bacterial (Infections and infestations) | 0 | 0 | 4 | 1 | 0 | 0 | 0 | 0 | 0
Pneumonia haemophilus (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia influenzal (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia moraxella (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia mycoplasmal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pneumonia parainfluenzae viral (Infections and infestations) | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia pseudomonal (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia respiratory syncytial viral (Infections and infestations) | 1 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Pneumonia serratia (Infections and infestations) | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia streptococcal (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pneumonia viral (Infections and infestations) | 0 | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 1
Postoperative wound infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Pseudomonas bronchitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pseudomonas infection (Infections and infestations) | 0 | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Pulpitis dental (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pyuria (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 0 | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory syncytial virus infection (Infections and infestations) | 1 | 1 | 12 | 1 | 0 | 0 | 0 | 4 | 3
Respiratory tract infection (Infections and infestations) | 0 | 2 | 8 | 0 | 0 | 0 | 0 | 0 | 1
Respiratory tract infection viral (Infections and infestations) | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rhinovirus infection (Infections and infestations) | 0 | 5 | 5 | 0 | 0 | 1 | 0 | 2 | 0
Rotavirus infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Staphylococcal bacteraemia (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Staphylococcal infection (Infections and infestations) | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Stenotrophomonas infection (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Stoma site infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Subcutaneous abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tracheitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 3 | 5 | 0 | 0 | 0 | 0 | 1 | 2
Urinary tract infection (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Varicella (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Viral infection (Infections and infestations) | 2 | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Viral pericarditis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Viral upper respiratory tract infection (Infections and infestations) | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Accident (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Face injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 1 | 1 | 0 | 0 | 1 | 3
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 2 | 3
Foreign body aspiration (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Foreign body in respiratory tract (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal procedural complication (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal stoma complication (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gastrostomy tube site complication (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Musculoskeletal procedural complication (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neurological procedural complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Post lumbar puncture syndrome (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 4
Post procedural complication (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Postoperative ileus (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Procedural dizziness (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Respiratory tract procedural complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Unintentional medical device removal (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Blood culture positive (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Coronavirus test positive (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Enterovirus test positive (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Human rhinovirus test positive (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oxygen saturation decreased (Investigations) | 0 | 4 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory rate increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory syncytial virus test positive (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rubulavirus test positive (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 2 | 3 | 2 | 0 | 1 | 0 | 0 | 1
Failure to thrive (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Feeding intolerance (Metabolism and nutrition disorders) | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ketoacidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Malnutrition (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Hip deformity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0
Joint contracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Kyphoscoliosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 4 | 0 | 0 | 0 | 0 | 1 | 2
Neuromuscular scoliosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Retrognathia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Scoliosis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 10 | 3 | 2 | 6 | 0 | 11 | 22
Brain stem glioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hair follicle tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Altered state of consciousness (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Brain hypoxia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Seizure (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Status epilepticus (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Device failure (Product Issues) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Device malfunction (Product Issues) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Device mechanical issue (Product Issues) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Urinary retention (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Testicular torsion (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 | 9 | 15 | 2 | 0 | 2 | 0 | 3 | 1
Adenoidal hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Apnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 5 | 0 | 0 | 0 | 0 | 0 | 2
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Bronchial secretion retention (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Obstructive sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 2 | 5 | 9 | 1 | 0 | 0 | 0 | 1 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 9 | 0 | 0 | 0 | 0 | 1 | 1
Respiratory symptom (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Positive airway pressure therapy (Surgical and medical procedures) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypovolaemic shock (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Infantile SMA Onset CS3A (N=13) | Infantile SMA Onset CS3B Previous Control (N=24) | Infantile SMA Onset CS3B Previous ISIS 396443 (N=65) | Infantile SMA Onset 232SM202 (N=12) | Later SMA Onset 232SM202 (N=8) | Later SMA Onset CS12 Type 2 (N=20) | Later SMA Onset CS12 Type 3 (N=25) | Later SMA Onset CS4 Previous Control (N=42) | Later SMA Onset CS4 Previous ISIS 396443 (N=83)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 6 | 1 | 1 | 2 | 0 | 1 | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 2 | 2 | 0 | 0 | 0 | 0 | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0 | 3 | 0 | 0 | 0 | 0 | 1 | 2
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Thrombocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Bradycardia (Cardiac disorders) | 1 | 0 | 6 | 1 | 0 | 0 | 0 | 1 | 0
Pericardial effusion (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Right atrial enlargement (Cardiac disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Right ventricular hypertrophy (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 2 | 4 | 5 | 1 | 0 | 0 | 0 | 1 | 2
Cryptorchism (Congenital, familial and genetic disorders) | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Developmental hip dysplasia (Congenital, familial and genetic disorders) | 1 | 1 | 3 | 1 | 1 | 1 | 0 | 1 | 5
High arched palate (Congenital, familial and genetic disorders) | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cerumen impaction (Ear and labyrinth disorders) | 2 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Ear pain (Ear and labyrinth disorders) | 1 | 0 | 2 | 0 | 0 | 0 | 2 | 0 | 4
Hyperacusis (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Motion sickness (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1
Myringosclerosis (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Precocious puberty (Endocrine disorders) | 0 | 2 | 4 | 0 | 0 | 1 | 0 | 1 | 0
Amblyopia (Eye disorders) | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Astigmatism (Eye disorders) | 1 | 2 | 3 | 0 | 1 | 0 | 1 | 0 | 1
Chalazion (Eye disorders) | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Eyelid cyst (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypermetropia (Eye disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Myopia (Eye disorders) | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 3 | 4
Strabismus (Eye disorders) | 0 | 1 | 4 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 4 | 1 | 0 | 0 | 0 | 2 | 2
Abdominal pain (Gastrointestinal disorders) | 2 | 1 | 4 | 1 | 0 | 0 | 1 | 3 | 7
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 3 | 5
Colitis ulcerative (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 3 | 7 | 22 | 1 | 3 | 1 | 1 | 9 | 11
Diarrhoea (Gastrointestinal disorders) | 4 | 8 | 16 | 2 | 2 | 1 | 0 | 6 | 11
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 2 | 5 | 0 | 0 | 1 | 0 | 2 | 0
Gastritis (Gastrointestinal disorders) | 1 | 1 | 2 | 0 | 0 | 0 | 1 | 0 | 2
Gastritis haemorrhagic (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 5 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal motility disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 4 | 9 | 0 | 0 | 1 | 0 | 0 | 1
Hiatus hernia (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Ileus paralytic (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Impaired gastric emptying (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lip dry (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lip swelling (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 1 | 6 | 0 | 0 | 2 | 2 | 8 | 15
Oral pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Saliva discolouration (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Salivary hypersecretion (Gastrointestinal disorders) | 1 | 6 | 10 | 0 | 0 | 0 | 0 | 0 | 1
Scalloped tongue (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Teething (Gastrointestinal disorders) | 0 | 4 | 9 | 0 | 0 | 0 | 0 | 0 | 0
Tooth impacted (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 7 | 9 | 23 | 3 | 4 | 7 | 4 | 18 | 35
Developmental delay (General disorders) | 0 | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 2 | 5 | 3 | 0 | 0 | 3 | 0 | 1
Gait disturbance (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0
Infusion site bruising (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Medical device site haemorrhage (General disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pain (General disorders) | 2 | 3 | 3 | 0 | 1 | 0 | 0 | 1 | 2
Peripheral swelling (General disorders) | 1 | 0 | 2 | 0 | 0 | 0 | 2 | 1 | 2
Pneumatosis (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 13 | 15 | 50 | 5 | 5 | 10 | 3 | 21 | 39
Hepatic steatosis (Hepatobiliary disorders) | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 2 | 1 | 0 | 0 | 1 | 0 | 1 | 2
Multiple allergies (Immune system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Seasonal allergy (Immune system disorders) | 0 | 3 | 9 | 0 | 0 | 1 | 2 | 3 | 5
Abdominal abscess (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Acute sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Adenovirus infection (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Bacterial disease carrier (Infections and infestations) | 0 | 4 | 4 | 0 | 0 | 0 | 0 | 0 | 1
Bacterial infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Bronchiolitis (Infections and infestations) | 2 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 1 | 10 | 2 | 1 | 2 | 0 | 7 | 5
Cellulitis (Infections and infestations) | 0 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Clostridium difficile infection (Infections and infestations) | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Conjunctivitis (Infections and infestations) | 2 | 3 | 8 | 0 | 0 | 0 | 0 | 1 | 4
Coronavirus infection (Infections and infestations) | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Covid-19 (Infections and infestations) | 4 | 1 | 16 | 5 | 2 | 4 | 5 | 8 | 16
Coxsackie viral infection (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Croup infectious (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cystitis (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 3
Ear infection (Infections and infestations) | 2 | 3 | 21 | 2 | 1 | 3 | 1 | 5 | 14
Ear infection fungal (Infections and infestations) | 0 | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Enterovirus infection (Infections and infestations) | 0 | 4 | 4 | 1 | 0 | 0 | 0 | 1 | 2
Eye infection (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fungal skin infection (Infections and infestations) | 0 | 1 | 2 | 0 | 0 | 1 | 0 | 1 | 0
Gastritis viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 2 | 9 | 2 | 1 | 3 | 0 | 4 | 11
Gastroenteritis viral (Infections and infestations) | 0 | 1 | 4 | 1 | 1 | 7 | 5 | 5 | 3
Gastrointestinal viral infection (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 1
Hand-foot-and-mouth disease (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3
Hordeolum (Infections and infestations) | 0 | 2 | 4 | 1 | 0 | 0 | 0 | 1 | 2
Impetigo (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 1 | 1
Influenza (Infections and infestations) | 2 | 3 | 13 | 0 | 1 | 4 | 3 | 6 | 16
Klebsiella infection (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 3 | 4 | 0 | 1 | 0 | 0 | 0 | 3
Lower respiratory tract infection viral (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Metapneumovirus infection (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Moraxella infection (Infections and infestations) | 0 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Mycoplasma infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 4 | 5 | 26 | 4 | 1 | 4 | 8 | 13 | 27
Oral candidiasis (Infections and infestations) | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Oral fungal infection (Infections and infestations) | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Otitis externa (Infections and infestations) | 1 | 0 | 4 | 1 | 0 | 0 | 0 | 0 | 3
Otitis media (Infections and infestations) | 4 | 4 | 14 | 1 | 1 | 4 | 0 | 5 | 6
Otitis media acute (Infections and infestations) | 2 | 2 | 3 | 0 | 0 | 0 | 0 | 2 | 2
Parainfluenzae virus infection (Infections and infestations) | 2 | 0 | 5 | 0 | 0 | 0 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 2 | 4 | 0 | 0 | 1 | 0 | 4 | 3
Pharyngitis streptococcal (Infections and infestations) | 1 | 0 | 2 | 0 | 1 | 3 | 3 | 4 | 8
Pneumonia (Infections and infestations) | 4 | 6 | 18 | 4 | 1 | 1 | 0 | 6 | 11
Pneumonia aspiration (Infections and infestations) | 0 | 2 | 7 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia bacterial (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1
Postoperative wound infection (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 1
Pseudomonas infection (Infections and infestations) | 0 | 6 | 11 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory syncytial virus infection (Infections and infestations) | 2 | 2 | 8 | 0 | 1 | 0 | 0 | 2 | 1
Respiratory tract infection (Infections and infestations) | 4 | 2 | 22 | 1 | 2 | 0 | 0 | 3 | 8
Respiratory tract infection bacterial (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory tract infection viral (Infections and infestations) | 2 | 1 | 6 | 0 | 2 | 2 | 0 | 1 | 2
Rhinitis (Infections and infestations) | 0 | 6 | 5 | 1 | 0 | 0 | 0 | 3 | 8
Rhinovirus infection (Infections and infestations) | 0 | 0 | 12 | 2 | 0 | 1 | 0 | 3 | 3
Serratia infection (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 1 | 2 | 6 | 2 | 0 | 2 | 0 | 3 | 6
Staphylococcal infection (Infections and infestations) | 0 | 1 | 7 | 1 | 0 | 0 | 0 | 0 | 0
Stenotrophomonas infection (Infections and infestations) | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Stoma site cellulitis (Infections and infestations) | 0 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Stoma site infection (Infections and infestations) | 1 | 1 | 4 | 0 | 0 | 0 | 0 | 0 | 0
Suspected covid-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tonsillitis (Infections and infestations) | 1 | 1 | 1 | 0 | 0 | 0 | 1 | 3 | 6
Tooth abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tracheitis (Infections and infestations) | 0 | 4 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 11 | 14 | 34 | 3 | 6 | 8 | 5 | 21 | 33
Upper respiratory tract infection bacterial (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 3 | 3 | 10 | 1 | 1 | 2 | 1 | 4 | 7
Viral infection (Infections and infestations) | 1 | 1 | 3 | 0 | 1 | 0 | 4 | 2 | 10
Viral upper respiratory tract infection (Infections and infestations) | 2 | 1 | 5 | 0 | 0 | 3 | 2 | 4 | 4
Accident (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 2 | 1
Anaesthetic complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1
Anaesthetic complication neurological (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 2 | 1 | 3 | 0 | 0 | 0 | 0 | 2 | 3
Concussion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 1 | 2 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 6
Endotracheal intubation complication (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0
Extraskeletal ossification (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 3 | 6 | 0 | 0 | 3 | 6 | 9 | 19
Femur fracture (Injury, poisoning and procedural complications) | 2 | 3 | 5 | 1 | 2 | 1 | 0 | 5 | 8
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Gastrointestinal stoma complication (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 3 | 1 | 1 | 0 | 0 | 0 | 0 | 2 | 3
Immunisation reaction (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1
Incision site swelling (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 1 | 7 | 0 | 0 | 2 | 0 | 3 | 3
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1 | 1 | 5 | 1 | 4
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 0
Palate injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Post lumbar puncture syndrome (Injury, poisoning and procedural complications) | 2 | 4 | 4 | 0 | 2 | 13 | 15 | 7 | 21
Post procedural complication (Injury, poisoning and procedural complications) | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 2
Post procedural constipation (Injury, poisoning and procedural complications) | 0 | 0 | 5 | 0 | 0 | 0 | 0 | 0 | 0
Post procedural contusion (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 1 | 3 | 0 | 0 | 0 | 1 | 1 | 0
Post procedural inflammation (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Procedural hypotension (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 5 | 5 | 15 | 2 | 2 | 6 | 11 | 19 | 29
Procedural pneumothorax (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Procedural vomiting (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 3
Respiratory tract procedural complication (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 1
Skin abrasion (Injury, poisoning and procedural complications) | 1 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 1
Stoma site discharge (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Stoma site erythema (Injury, poisoning and procedural complications) | 0 | 1 | 2 | 1 | 0 | 0 | 0 | 0 | 0
Stoma site haemorrhage (Injury, poisoning and procedural complications) | 0 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Stoma site hypergranulation (Injury, poisoning and procedural complications) | 0 | 4 | 5 | 0 | 0 | 0 | 0 | 0 | 0
Suture rupture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 0 | 2 | 0 | 0 | 1 | 0 | 2 | 4
Tooth fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 3
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Wound secretion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Activated partial thromboplastin time prolonged (Investigations) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2
Blood albumin decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blood iron decreased (Investigations) | 0 | 0 | 3 | 1 | 0 | 0 | 0 | 0 | 0
Blood potassium decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Bone density decreased (Investigations) | 1 | 1 | 1 | 0 | 0 | 1 | 0 | 3 | 1
Breath sounds abnormal (Investigations) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Cardiac murmur (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Clostridium test positive (Investigations) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Crystal urine present (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 6
Electrocardiogram qt prolonged (Investigations) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 2 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Haemoglobin decreased (Investigations) | 0 | 1 | 2 | 1 | 0 | 0 | 0 | 0 | 0
Heart rate increased (Investigations) | 3 | 2 | 4 | 3 | 0 | 0 | 0 | 2 | 0
Mean platelet volume decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Occult blood positive (Investigations) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Oxygen consumption decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Oxygen saturation decreased (Investigations) | 1 | 7 | 18 | 2 | 0 | 0 | 1 | 2 | 3
Platelet count increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Prothrombin time prolonged (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pseudomonas test positive (Investigations) | 0 | 1 | 6 | 0 | 0 | 0 | 0 | 0 | 0
Qrs axis abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Red blood cell count increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Red blood cell sedimentation rate increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Sars-cov-2 test positive (Investigations) | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 1
Vitamin d decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1
Von willebrand's factor activity decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Weight decreased (Investigations) | 0 | 0 | 3 | 1 | 0 | 0 | 1 | 1 | 3
Weight increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 0
White blood cell count increased (Investigations) | 0 | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 0
White blood cells urine positive (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 2 | 6 | 1 | 0 | 1 | 1 | 4 | 2
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1
Feeding intolerance (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypochloraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 3 | 0 | 0 | 0 | 0 | 1 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 3 | 10 | 0 | 0 | 0 | 0 | 1 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Iron deficiency (Metabolism and nutrition disorders) | 0 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Malnutrition (Metabolism and nutrition disorders) | 1 | 0 | 6 | 0 | 0 | 0 | 0 | 0 | 4
Metabolic acidosis (Metabolism and nutrition disorders) | 2 | 1 | 2 | 0 | 0 | 0 | 0 | 2 | 2
Metabolic alkalosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Obesity (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 2 | 4
Vitamin d deficiency (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 1 | 1
Weight gain poor (Metabolism and nutrition disorders) | 1 | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 3 | 4 | 2 | 0 | 3 | 3 | 5 | 6
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 7 | 2 | 1 | 3 | 11 | 11 | 15
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0
Deformity thorax (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 3
Hip deformity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 9 | 0 | 2 | 2 | 0 | 1 | 2
Joint contracture (Musculoskeletal and connective tissue disorders) | 4 | 6 | 16 | 2 | 1 | 8 | 3 | 11 | 21
Joint laxity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 | 2 | 2 | 0 | 0 | 0 | 0 | 1 | 2
Knee deformity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Kyphoscoliosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 5 | 0 | 0 | 0 | 0 | 1 | 3
Kyphosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 10 | 0 | 1 | 1 | 1 | 2 | 3
Limb asymmetry (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Muscle atrophy (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscle contracture (Musculoskeletal and connective tissue disorders) | 5 | 6 | 18 | 2 | 1 | 6 | 1 | 17 | 37
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3 | 1 | 0 | 1 | 0 | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Neuromuscular scoliosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 1
Osteopenia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 9 | 0 | 0 | 2 | 0 | 1 | 3
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 7 | 0 | 2 | 2 | 0 | 2 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 4 | 7 | 1 | 1 | 1 | 6 | 4 | 6
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Scoliosis (Musculoskeletal and connective tissue disorders) | 6 | 10 | 38 | 3 | 5 | 6 | 2 | 22 | 33
Spinal deformity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tendinous contracture (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 2
Hair follicle tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 1
Areflexia (Nervous system disorders) | 2 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 1
Autonomic nervous system imbalance (Nervous system disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cognitive disorder (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Disturbance in attention (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 1 | 2
Dysarthria (Nervous system disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 4 | 3 | 8 | 1 | 3 | 5 | 17 | 20 | 24
Horner's syndrome (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hyporeflexia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Intracranial pressure increased (Nervous system disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Lethargy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1
Migraine (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 1
Motor developmental delay (Nervous system disorders) | 3 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 1
Muscle contractions involuntary (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 1 | 4
Myoclonus (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nystagmus (Nervous system disorders) | 0 | 0 | 4 | 1 | 0 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1
Tremor (Nervous system disorders) | 1 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 3
Device dislocation (Product Issues) | 1 | 0 | 5 | 0 | 0 | 1 | 0 | 0 | 0
Device malfunction (Product Issues) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Agitation (Psychiatric disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 2 | 2 | 0 | 3 | 3 | 1 | 4
Anxiety disorder (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Attention deficit hyperactivity disorder (Psychiatric disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 1 | 1 | 1
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Encopresis (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Irritability (Psychiatric disorders) | 0 | 2 | 4 | 0 | 0 | 0 | 0 | 0 | 1
Learning disability (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mental status changes (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Panic attack (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Kidney enlargement (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 2
Pollakiuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 3
Proteinuria (Renal and urinary disorders) | 0 | 1 | 7 | 1 | 0 | 0 | 2 | 2 | 8
Urinary retention (Renal and urinary disorders) | 1 | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 1
Heavy menstrual bleeding (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Testicular atrophy (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 4 | 1 | 0 | 0 | 0 | 0 | 1
Adenoidal hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 3 | 0 | 0 | 1 | 0 | 0 | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 5 | 1 | 0 | 0 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 5 | 2 | 9 | 1 | 0 | 0 | 0 | 0 | 2
Bronchial wall thickening (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 4 | 16 | 5 | 5 | 6 | 2 | 15 | 29
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 3 | 2 | 0 | 0 | 0 | 0 | 1
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Epiglottic oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 11 | 0 | 0 | 0 | 3 | 1 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 4 | 0 | 0 | 1 | 0 | 0 | 2
Increased bronchial secretion (Respiratory, thoracic and mediastinal disorders) | 2 | 4 | 8 | 0 | 0 | 0 | 0 | 0 | 1
Increased upper airway secretion (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 6 | 0 | 0 | 0 | 0 | 0 | 1
Increased viscosity of upper respiratory secretion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Laryngospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Lower respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 1
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 6 | 2 | 0 | 1 | 0 | 1 | 9
Noninfective bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Obstructive sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 0 | 2 | 0 | 4 | 5
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 3 | 1 | 1 | 4 | 3 | 8 | 12
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 3 | 0 | 0 | 0 | 1 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3 | 0 | 0 | 1 | 0 | 2 | 5
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Rales (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 3 | 1 | 1 | 0 | 1 | 0 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 5 | 5 | 1 | 0 | 0 | 0 | 0 | 1
Restrictive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 1 | 2
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 1 | 0 | 1 | 0 | 0 | 3 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 7 | 1 | 2 | 1 | 1 | 4 | 8
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1
Sputum discoloured (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 4 | 0 | 0 | 0 | 1 | 1 | 3
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 2 | 1
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blister (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 2 | 3 | 0 | 0 | 0 | 0 | 0 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 3 | 3 | 0 | 0 | 1 | 0 | 0 | 4
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 0 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2
Eczema (Skin and subcutaneous tissue disorders) | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 4 | 2
Erythema (Skin and subcutaneous tissue disorders) | 1 | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Keratosis pilaris (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Miliaria (Skin and subcutaneous tissue disorders) | 0 | 3 | 2 | 0 | 0 | 1 | 0 | 1 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3
Rash (Skin and subcutaneous tissue disorders) | 1 | 4 | 7 | 0 | 0 | 2 | 0 | 6 | 8
Scab (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Skin mass (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 2 | 2 | 0 | 0 | 0 | 0 | 3 | 6
Hypertension (Vascular disorders) | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 3 | 1 | 0 | 1 | 0 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Our agreement is subject to confidentiality but generally the PI can publish, for noncommercial purposes only, results and methods of the trial, but no other Sponsor Confidential Information. PI must give Sponsor no less than 60 days to review any manuscript for a proposed publication and must delay publication for up to an additional 90 days thereafter if Sponsor needs to file any patent application to protect any of Sponsor's intellectual property contained in the proposed publication.

DOCUMENTS (2):
  • Study Protocol (2021-10-20): https://cdn.clinicaltrials.gov/large-docs/24/NCT02594124/Prot_000.pdf
  • Statistical Analysis Plan (2023-09-06): https://cdn.clinicaltrials.gov/large-docs/24/NCT02594124/SAP_001.pdf